CLINICAL TRIAL: NCT02727218
Title: Effectiveness and Safety of Early Removal of Chest Tubes After Thoracoscopic Lung Resection and Biopsies ; a Prospective Randomized Controlled Study.
Brief Title: Safety of Early Removal of Chest Tubes After Thoracoscopic Lung Biopsies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, KATZ AMIT M.D., Dr, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0361-15rmb
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Non-Neoplastic Thoracic Disorder; Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chest tube removal after 3 hours (Experimental): 30 patients, post thoracoscopic lobectomy, segmentectomy, thoracoscopic mediastinal biopsy, will undergo chest tube removal after 3 hours.
  Interventions: Procedure: Chest tube removal
- delayed chest tube removal (Active Comparator): 30 patients, post thoracoscopic lobectomy, segmentectomy, thoracoscopic mediastinal biopsy, will undergo chest tube removal according to the department's protocol, most probably post operative day 1 (POD1)
  Interventions: Procedure: Chest tube removal

INTERVENTIONS:
Procedure: Chest tube removal — chest tube removal post thoracoscopic surgery

SUMMARY:
prospective study, involves 60 patients underwent thoracoscopic surgery, the patients will be divided into two groups, the first group will undergo early chest tube removal - after three hours, the second group will have late chest tube removal according to the department's protocol.

the study aims to prove the possibility and non inferiority for early chest tube removal for thoracoscopic surgeries with non complicated surgical course.

DETAILED DESCRIPTION:
Presence of chest tube post thoracoscopic surgery is associated with increased morbidities like wound infection, pain, and prolong the hospital admission Corse, in the other hand, early chest tube removal is associated with increased the need for recurrent active intervention like pleural tapping for re-accumulated pleural effusion.

Method: randomized prospective study includes 60 patients who underwent thoracoscopic lobectomy/segmentectomy/ thoracoscopic mediastinal biopsy.

The study will exclude patients with difficult operative course ( intraoperative finding of significant adhesions/ intraoperative injury of the lung parenchyma/ intraoperative bleeding/failure of extubation ) and patient with post operative findings of ( bleeding in the chest tube more than 100 ml in the first hour, persistent air leak, non expanded lung on chest x-ray ) The patients will be divided into two groups, the first group - 30 patients - will undergo chest tube removal after three hours, and the second group will undergo chest tube removal according to the treating department protocol.

All patients will be evaluated regarding the pain level - subjective and objective -, admission period, infection, and the need for invasive intervention.

The patients will be evaluated during the admission, after one week and after two weeks.

ELIGIBILITY:
Inclusion Criteria:

* patient's who undergo thoracoscopic lung resection ( lobectomy or segmentectomy ), or thoracoscopic mediastinal biopsy.
* post op there was no bleeding, the lung expanded, no persistent air leak, fluid discharge in the chest tube less than 100 ml, the patient underwent extubation.
* patients with who read and signed informed consent regarding the participation of the study.

Exclusion Criteria:

* Patients who underwent thoracoscopic segmental resection due to primary spontaneous pneumothorax.
* patients who underwent thoracoscopic pleural biopsy for possible malignancy.
* patients under 18 year old.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Non complicated early chest tube removal | two weeks
  the patient with inclusion criteria can undergo early chest tube removal after three hours with no need for chest tube insertion, or pleural tapping for recurrent pleural effusion,
Complicated early chest tube removal | two weeks
  Patients who underwent early chest tube removal 3 hours after surgery are more liable for reinsertion of chest tube or active pleural tapping.

CONTACTS AND LOCATIONS:
Overall Officials: Ran Kremer, MD, Study Director — Rambam Health Care Campus

REFERENCES:
- [Background] Chang AC, Yee J, Orringer MB, Iannettoni MD. Diagnostic thoracoscopic lung biopsy: an outpatient experience. Ann Thorac Surg. 2002 Dec;74(6):1942-6; discussion 1946-7. doi: 10.1016/s0003-4975(02)04164-4. PMID 12643377
- [Background] Gomez-Caro A, Roca MJ, Torres J, Cascales P, Terol E, Castaner J, Pinero A, Parrilla P. Successful use of a single chest drain postlobectomy instead of two classical drains: a randomized study. Eur J Cardiothorac Surg. 2006 Apr;29(4):562-6. doi: 10.1016/j.ejcts.2006.01.019. Epub 2006 Feb 21. PMID 16495069
- [Background] Okur E, Baysungur V, Tezel C, Sevilgen G, Ergene G, Gokce M, Halezeroglu S. Comparison of the single or double chest tube applications after pulmonary lobectomies. Eur J Cardiothorac Surg. 2009 Jan;35(1):32-5; discussion 35-6. doi: 10.1016/j.ejcts.2008.09.009. Epub 2008 Oct 16. PMID 18929492
- [Background] Younes RN, Gross JL, Aguiar S, Haddad FJ, Deheinzelin D. When to remove a chest tube? A randomized study with subsequent prospective consecutive validation. J Am Coll Surg. 2002 Nov;195(5):658-62. doi: 10.1016/s1072-7515(02)01332-7. PMID 12437253
- [Background] Refai M, Brunelli A, Salati M, Xiume F, Pompili C, Sabbatini A. The impact of chest tube removal on pain and pulmonary function after pulmonary resection. Eur J Cardiothorac Surg. 2012 Apr;41(4):820-2; discussion 823. doi: 10.1093/ejcts/ezr126. Epub 2011 Dec 21. PMID 22219425
- [Background] Yu H. Management of pleural effusion, empyema, and lung abscess. Semin Intervent Radiol. 2011 Mar;28(1):75-86. doi: 10.1055/s-0031-1273942. PMID 22379278
- [Background] Bjerregaard LS, Jensen K, Petersen RH, Hansen HJ. Early chest tube removal after video-assisted thoracic surgery lobectomy with serous fluid production up to 500 ml/day. Eur J Cardiothorac Surg. 2014 Feb;45(2):241-6. doi: 10.1093/ejcts/ezt376. Epub 2013 Jul 19. PMID 23872457
- [Background] McKenna RJ Jr, Mahtabifard A, Pickens A, Kusuanco D, Fuller CB. Fast-tracking after video-assisted thoracoscopic surgery lobectomy, segmentectomy, and pneumonectomy. Ann Thorac Surg. 2007 Nov;84(5):1663-7; discussion 1667-8. doi: 10.1016/j.athoracsur.2007.05.058. PMID 17954081
- [Background] Cerfolio RJ, Bryant AS. Results of a prospective algorithm to remove chest tubes after pulmonary resection with high output. J Thorac Cardiovasc Surg. 2008 Feb;135(2):269-73. doi: 10.1016/j.jtcvs.2007.08.066. PMID 18242249
- [Background] Nakanishi R, Fujino Y, Yamashita T, Oka S. A prospective study of the association between drainage volume within 24 hours after thoracoscopic lobectomy and postoperative morbidity. J Thorac Cardiovasc Surg. 2009 Jun;137(6):1394-9. doi: 10.1016/j.jtcvs.2008.10.035. Epub 2009 Mar 9. PMID 19464455
- [Background] Gottgens KW, Siebenga J, Belgers EH, van Huijstee PJ, Bollen EC. Early removal of the chest tube after complete video-assisted thoracoscopic lobectomies. Eur J Cardiothorac Surg. 2011 Apr;39(4):575-8. doi: 10.1016/j.ejcts.2010.08.002. Epub 2010 Sep 15. PMID 20833554